CLINICAL TRIAL: NCT03509558
Title: Transcutaneous Spinal Stimulation With Intensive Physical Therapy for Locomotion
Brief Title: Transcutaneous Spinal Stimulation and Exercise for Locomotion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Chet Moritz, Associate Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003070
Record Dates: First submitted 2018-03-24; First posted 2018-04-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal electrical stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcutaneous spinal stimulation & Physical therapy (Active Comparator): Transcutaneous electrical stimulation combined with physical therapy that targets rehabilitation of walking and standing functions
  Interventions: Device: Transcutaneous spinal stimulation; Other: Physical Therapy
- Physical therapy only (Active Comparator): Physical therapy that targets rehabilitation of walking and standing functions
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: Transcutaneous spinal stimulation — Non-invasive electrical stimulation of spinal cord over the skin combined with physical therapy to improve walking and standing functions
  Other Names: Physical Therapy
  Arms: Transcutaneous spinal stimulation & Physical therapy
Other: Physical Therapy — physical therapy to improve walking and standing functions

SUMMARY:
Growing evidence indicates that electrical spinal cord stimulation improves motor functions both immediately and over the long term via modulating the excitability of spinal circuitry in patients with spinal cord injury. Recently, a novel, non-invasive, well-tolerated, and painless lumbosacral transcutaneous electrical stimulation strategy was demonstrated to be effective in improving lower limb motor function in participants with spinal cord injury. Our current project, cervical transcutaneous electrical stimulation and intensive exercise for arms and hands are also revealing a significant improvement in upper extremity function. Additionally, the subject and caregiver noted that stair climbing ability has been substantially enhanced starting from the first week of cervical stimulation treatment and continues to date.

This study is a prospective efficacy trial of combined transcutaneous cervical and lumbosacral electrical stimulation with physical therapy for improving locomotion in people with anatomically incomplete tetraplegia and paraplegia.

This experiment design consists of testing walking function with and without transcutaneous spinal cord stimulation. A two to four-phase intervention program will include physical therapy and spinal cord stimulation with physical therapy. The length of any intervention phase, and number of measurements performed during that phase, will be determined by multiple factors, including participants' health condition, availability, and response to intervention. Between each intervention, washout periods of up to one month may be used to determine any after-effects of the interventions.

The intervention arms will be repeated if the functional improvement does not reach a plateau during the first two months of intervention. Physical therapy will include functional training (e.g., walking training) and strength training. Each spinal cord stimulation with physical therapy intervention block can use transcutaneous lumbosacral stimulation or cervical and lumbosacral stimulation. Both immediate and lasting improvements in lower extremity function and autonomic function via transcutaneous spinal cord stimulation and intensive physical therapy may be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Has spinal cord injury (T12 or higher level) of at least 1-year duration
* Is between 21 and 70 years of age
* Has difficulty with leg functions and mobility in activities of daily living (e.g. walking, transferring surface to surface, standing)
* Has stable medical condition without cardiopulmonary disease or frequent autonomic dysreflexia that would contraindicate participation in lower extremity rehabilitation or testing activities
* Is capable of performing simple cued motor tasks
* Has ability to attend up to 5 sessions per week physical therapy sessions and testing activities
* Has adequate social support to be able to participate in training and assessment sessions, up to 5 sessions per week, for the duration of up to 11 months within the study period
* Is volunteering to be involved in this study
* Cleared for gait training by the primary physician of the subject
* Has the ability to read and speak English

Exclusion Criteria:

* Has autoimmune etiology of spinal cord dysfunction/injury
* Has history of additional neurologic disease, such as stroke, multiple sclerosis, traumatic brain injury, etc.
* Has peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy, etc.)
* Has rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
* Has significant medical disease; including uncontrolled systemic hypertension with values above 170/100 mmHg; cardiac or pulmonary disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation.
* Has active cancer
* Has cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention
* Has unhealed fracture, contracture, pressure sore, urinary tract infection, or other illnesses that might interfere with lower extremity rehabilitation or testing activities
* Has any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician
* is pregnant
* is dependent on ventilation support
* Has implanted stimulator (e.g. epidural stimulator, vagus nerve stimulator, pacemaker, cochlear implant, etc)
* Has depression or anxiety based on the Center for Epidemiologic Studies Depression Scale (CESD) (score >16/60) and General Anxiety Disorder-7 item Questionnaire (score >9/21), respectively
* Has alcohol and/or drug abuse
* Has cognitive impairment based on Short Portable Mental Status Questionnaire (SPMSQ) (score >2/10)
* is unable to read and/or comprehend the consent form
* is unable to understand the instructions given as part of the study
* Has established osteoporosis and taking medication for osteoporosis treatment
* Has bone mineral density T scores ≤ -3.5 or Z scores ≤ -2.5 in the anteroposterior lumbar spine and/or proximal femur measured by a DEXA scan for subjects weight bearing and ambulating outside of a body-weight supporting exoskeleton (if participants are clear for other criteria and have not been examined by Dual Energy Xray Absorptiometry (DEXA) at the screening, we will ask participants to undergo DEXA to reveal any risk of weight bearing activity)
* Has low-energy fracture history before or after spinal cord injury
* History of orthopedic surgery in lower extremities that may be a confounding factor for interpretation of the results (such as tendon transfer, tendon or muscle lengthening for spasticity management, arthrodesis, etc.)
* fixed lower extremity joint contractures
* is taller than 80 inches and/or more than 350 pounds body weights, due to the limitation of the experimental equipment such as the body weight support system
* lacks the ability to fully comprehend and/or perform study procedures in the investigator's opinion/judgement
* has history of severe allergy (i.e. allergic reaction that could not be treated with antihistaminic medication)
* has malabrosption syndrome, primary hyperthyroidism, and/or hypogonadism
* has a history of seizures
* has chronic headaches or migraines
* has deep brain stimulators, metallic devices in the head such as aneurysm clips/coils and stents, vagus nerve stimulators

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test | 1-11 months
  Measurement of walking ability. The distance is reported in meter.
Two-minute walk test | 1-11 months
  A measurement of endurance that assesses walking distance over two minutes.

SECONDARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Examination | 1-11 months
  Standard neurologic examination that is routinely used to determine the levels and severity of spinal cord injury. Includes manual muscle strength testing and dermatomal light touch and pin prick sensory examination.
Somatosensory evoked potentials | 1-11 months
  Measurement of latency of electrical potentials that is recorded by surface electrodes over the scalp following electrical stimulation of peripheral nerve from the wrist. The latency of the response is reported in micro-seconds.
Somatosensory evoked potentials | 1-11 months
  Measurement of amplitude of electrical potentials that is recorded by surface electrodes over the scalp following electrical stimulation of peripheral nerve from the wrist. The amplitude of the response is reported in micro-volts.
Motor evoked potentials | 1-11 months
  Measurement of latency of electrical potentials that is recorded by surface electrodes over the skin of limb muscles following spinal stimulation or magnetic stimulation of brain over the scalp. The latency of the response is reported in micro-seconds.
Motor evoked potentials | 1-11 months
  Measurement of amplitude of electrical potentials that is recorded by surface electrodes over the skin of limb muscles following spinal stimulation or magnetic stimulation of brain over the scalp. The amplitude of the response is reported in micro-volts.
Berg Balance Test | 1-11 months
  Measurement of balance in standing and sitting. The balance score consists of 14 items and is reported in the scale of 56 (each items are score in 0-4).
Ten-meter walk test | 1-11 months
  Measurement of walking ability. The walking speed is reported in meter per second.
Gait analysis | 1-11 months
  Measurement of leg function and walking ability. Joint angle is reported in degree angle. Step length is reported in centimeters and swing time is reported in seconds.
Kinetic and kinematic gait analysis using 3D camera system | 1-11 months
  Measurement of leg function and walking ability. Velocity is reported in meter per second.
Electromyography recording of lower extremity and trunk muscles | 1-11 months
  Measurement of muscle and nerve functions. The muscle activities are reported in micro-volts.
Spinal Cord Injury - Quality of Life (SCI-QOL) questionnaire | 1-11 months
  Patient reported quality of life scale. The SCI-QOL consists of 19 item banks, and is reported by T-score comparing the mean of the functional level in the population.
Spinal Cord Injury - Functional Index (SCI-FI) questionnaire | 1-11 months
  Patient reported functional scale. The SCI-QOL consists of 10 item banks, and is reported by T-score comparing the mean of the functional level in the population.
Modified Ashworth Scale | 1-11 months
  Measurement of spasticity. Tests resistance to passive movement about joints. Score range from 0-4, with 6 choices.
Neurogenic Bowel Dysfunction Score | 1-11 months
  self-report questionnaire designed to help healthcare professionals evaluate the effectiveness of their patient's current bowel management routine by assessing the impact it has on the patient's quality of life.
  Questions ask about background parameters (n=8), faecal incontinence (n=10), constipation (n=10), obstructed defecation (n=8), and impact on quality of life (QOL).
Neurogenic Bladder Symptom Score | 1-11 months
  objective and validated self-report questionnaire to assess bladder symptoms in patients with neurogenic bladder dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No